CLINICAL TRIAL: NCT04531605
Title: Feasibility and Acceptability of an Intervention to Optimize Retention in Care and Adherence to Anti-retroviral Therapy Amongst Adolescents Living With HIV in Rwanda
Brief Title: Optimizing Retention in Care and Adherence to Anti-retroviral Therapy Amongst Adolescents Living With HIV in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youth Development Labs, Inc dba YLabs (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 12-week program of combined life-skills training and financial incentives (YBank program) described in more detail below.
  1. Life-skills training: Every 4 weeks through the 12 week program, life-skills training sessions will be delivered during peer-group sessions at the clinic. Topics include economic empowerment, financial literacy, healthy relationships, and anti-retroviral therapy (ART) adherence.
  2. Financial incentives: The incentives program combines an immediate financial reward with a long-term savings opportunity. For clinic attendance, 500 RWF (~$0.50) will be deposited into participants' mobile money short-term account, where funds will be immediately accessible, and 1500 RWF (~$1.50) will be deposited into their savings account upon completing the program. If participants demonstrate a suppressed viral load at a clinic appointment, an additional 1000 RWF (~$1) will be deposited to their short-term account and 3000 RWF (~$3) into their saving account.
  Interventions: Behavioral: YBank program

INTERVENTIONS:
Behavioral: YBank program — Adolescents participated in a 12-week peer-led life skills trainings at clinics and received financial incentives via mobile money upon clinic attendance and demonstration of suppressed viral load.

SUMMARY:
HIV has now become the leading cause of death amongst adolescents in Africa with over 2.1 million adolescents (aged 10-19 years old) living with HIV today. Poor adherence to anti-retroviral therapy (ART) leads to suppressed immune function, treatment failure, increased morbidity and mortality with significant costs to households and health systems.

The investigators aim to undertake a feasibility study of an intervention targeting adolescents living with HIV in Rwanda built on two components.

1. Life-skills training: Adolescents receive training on economic empowerment, financial literacy, healthy relationships and adherence during the peer group sessions.
2. Financial incentives: Combined short-term and long-term incentives for clinic attendance and suppressed viral load that will be delivered through mobile banking.

DETAILED DESCRIPTION:
HIV has now become the leading cause of death amongst adolescents in Africa with over 2.1 million adolescents (aged 10-19 years old) living with HIV today. Increased mortality amongst HIV-infected adolescents is primarily caused by poor adherence to anti-retroviral therapy (ART). Adherence to ART is critical to suppress HIV viral load, sustain immune function, and avoid opportunistic infections and death. Poor adherence leads to suppressed immune function, treatment failure, increased morbidity and mortality with significant costs to households and health systems. In our clinic population in Rwanda, 29% of 12-19 years olds have a non-suppressed viral load due to poor adherence. These findings have been reflected in studies throughout the US, Europe and sub-Saharan Africa.

The evidence base for effective adherence interventions that successfully address the multiple barriers to adherence is very limited. Conditional cash transfers have shown promise as a potential strategy. The investigators aim to undertake a feasibility study of an intervention targeting adolescents living with HIV in Rwanda built on two components.

1. Life-skills training: Adolescents receive training on economic empowerment, financial literacy, healthy relationships and adherence during the peer group sessions.
2. Financial incentives: Combined short-term and long-term incentives for clinic attendance and suppressed viral load that will be delivered through mobile banking. On admission to the program adolescents are provided with a bank account. The rewards delivered to the adolescent are divided into a long-term and short term component. The long-term incentive accrues and can only be accessed on graduation from the program. The short-term component can be accessed immediately.

The aim of this preliminary study is not to assess for efficacy of the intervention (virological suppression and clinic attendance). This preliminary study aims to assess the feasibility of the program and data collection strategy in preparation for a large scale multi-center evaluation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adolescents 12 to 19-years-old who are aware of their HIV-positive serostatus
* Prescribed anti-retroviral therapy for more than 1 year
* Has given informed consent with full capacity to study participation (plus parent/guardian consent as all participants will be under 21 years)
* Enrolled in care at one of the study site

Exclusion Criteria:

* HIV-negative
* HIV-positive but not prescribed ART or on ART for less than 1 year
* Not enrolled in care at the HIV clinic; younger than 12 years and older than 19 years
* No parent or named guardian who is over the age of 19 years

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Experiences and views of adolescents, caregivers of participants, and health care professionals caring for participants of receiving the YBank intervention | 3 months
  Semi-structured interviews will be conducted with adolescents, caregivers and two health workers randomly selected from each site during and directly following the 12-week intervention period. Themes to be explored in the interviews include experiences with receiving incentives and attending trainings, the impact of the intervention on caregivers and adolescents, and how the incentives will be spent. Face-to-face interviews will be conducted in Kinyarwanda or French by trained interviewers.

IPD SHARING:
Plan to Share IPD: No